CLINICAL TRIAL: NCT04307693
Title: Randomized Controlled Clinical Trials of Lopinavir/Ritonavir or Hydroxychloroquine in Patients With Mild Coronavirus Disease (COVID-19)
Brief Title: Comparison of Lopinavir/Ritonavir or Hydroxychloroquine in Patients With Mild Coronavirus Disease (COVID-19)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early because no patients were further enrolled since mid-Apr 2020.
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Han Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2020-0472-0001
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Lopinavir; lopinavir-ritonavir drug combination; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Multicenter, open labelled, randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lopinavir/ritonavir (Experimental): Lopinavir/ritonavir 200mg/100mg 2 tablets by mouth, every 12 hours for 7-10 days
  Interventions: Drug: Lopinavir/ritonavir
- Hydroxychloroquine (Active Comparator): Hydroxychloroquine 400mg by mouth, every 24 hours for 7-10 days
  Interventions: Drug: Hydroxychloroquine sulfate
- Control (No Intervention): No lopinavir/ritonavir and hydroxychloroquine

INTERVENTIONS:
Drug: Lopinavir/ritonavir — Lopinavir / Ritonavir tablet
  Other Names: Kaletra
  Arms: Lopinavir/ritonavir
Drug: Hydroxychloroquine sulfate — Hydroxychloroquine sulfate tablet
  Other Names: Oxiklorin
  Arms: Hydroxychloroquine

SUMMARY:
In vitro studies revealed that lopinavir/ritonavir and hydroxychloroquine have antiviral activity against Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). However, there is no clinical studies on the reduction of viral load in patients with COVID-19. This study investigate whether lopinavir/ritonavir or hydroxychloroquine reduces viral load from respiratory specimen in patients with mild COVID-19.

DETAILED DESCRIPTION:
This multicenter study is an open-labelled, randomized clinical trial for 1:1:1 ratio of lopinavir/ritonavir, hydroxychloroquine, or control arm.

ELIGIBILITY:
Inclusion Criteria:

* confirmed mild COVID-19 (NEWS scoring system 0-4)

Exclusion Criteria:

* unable to take oral medication
* pregnancy or breast feeding
* immunocompromised patients
* creatinine clearance (CCL) < 30 mL/min
* aspartate transaminase (AST) or alanine transaminase (ALT) > 5 times Upper limit of normal (ULN)

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Viral load | hospital day 3, 5, 7, 10, 14, 18
  Area under the curve (AUC) of Ct value or viral copies number per mL

SECONDARY OUTCOMES:
Viral load change | hospital day 3, 5, 7, 10, 14, 18
  Viral load change (log10 viral load assessed by reverse transcription-PCR) during hospital day 3, 5, 7, 10, 14, 18)
Time to clinical improvement (TTCI) | up to 28 days
  Time to clinical improvement (TTCI) is defined as the time to normalization of fever, respiratory rate, and oxygen saturation, and alleviation of cough within at least 72 hours
Percentage of progression to supplemental oxygen requirement by day 7 | hospital day 7
  Percentage of progression to supplemental oxygen requirement by day 7
Time to NEWS2 (National Early Warning Score 2) of 3 or more maintained for 24 hours by day 7 | hospital day 7
  Time to NEWS2 (National Early Warning Score 2) of 3 or more maintained for 24 hours by day 7
Time to clinical failure, defined as the time to death, mechanical ventilation, or ICU admission | up to 28 days
  Time to clinical failure, defined as the time to death, mechanical ventilation, or ICU admission
Rate of switch to Lopinavir/ritonavir or hydroxychloroquine by day 7 | hospital day 7
  Rate of switch to Lopinavir/ritonavir or hydroxychloroquine by day 7
adverse effects | up to 28 days
  Safety and tolerability, as assessed by adverse effects
Concentration of Lopinavir/ritonavir and hydroxychloroquine | 1, 2, 4, 5, 12 hours after taking intervention medicine
  Concentration of Lopinavir/ritonavir and hydroxychloroquine

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lipsitch M, Perlman S, Waldor MK. Testing COVID-19 therapies to prevent progression of mild disease. Lancet Infect Dis. 2020 Dec;20(12):1367. doi: 10.1016/S1473-3099(20)30372-8. Epub 2020 May 6. No abstract available. PMID 32618282